CLINICAL TRIAL: NCT04141371
Title: Effect of Molar Sodium Lactate Filling on Cerebral Hemodynamics in Patients With Severe Meningeal Hemorrhage Multicenter Randomized Study
Brief Title: Molar Sodium Lactate Filling in Severe Meningeal Hemorrhage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19-PP-15
Record Dates: First submitted 2019-10-25; First posted 2019-10-28 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: paticipant and radiologists are masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Molar Sodium Lactate (Active Comparator)
  Interventions: Drug: Molar Sodium Lactate
- physiological serum (Placebo Comparator)
  Interventions: Drug: physiological serum

INTERVENTIONS:
Drug: Molar Sodium Lactate — daily 3-hour infusion of sodium molar lactate during the vasospasm period
  Arms: Molar Sodium Lactate
Drug: physiological serum — daily saline infusion over 3 hours during the vasospasm period
  Arms: physiological serum

SUMMARY:
Subarachnoid hemorrhage by aneurysmal rupture is a serious condition associated with a high mortality rate. Among the complications presented by these patients, vasospasm is one of the main causes of secondary aggravation, in particular the appearance of delayed neurological deficits following the induced cerebral ischemia. Classically occurring between the 4th and 12th day, with a peak on D7, its prevention is currently often ineffective.

In recent years, many studies have shown that sodium lactate could be an interesting product for neuroprotection. In addition to an anti-osmotic effect that has been demonstrated by our team in the context of post-traumatic intracranial hypertension, a metabolic action has also been observed in periods of metabolic attacks induced by brain attacks. Recently, a vasodilatory action of sodium lactate has been observed from an experimental and clinical point of view.

The purpose of this work is to observe the effect of sodium lactate, compared to placebo, on cerebral hemodynamics measured by perfusion CT (Mean Transit Time MTT) in a population of patients with hemorrhage under the arachnoid.

This work is the preliminary work of a study that will investigate the potential preventive protective effect of sodium lactate on the incidence of vasospasm.

ELIGIBILITY:
Inclusion Criteria:

* Any patient over 18 years of age with severe meningeal hemorrhage defined by a WFNS≥3 score will be included in the study.
* Treated by endovascular embolization or surgically within 48 hours
* After obtaining the informed consent of the patient, or his relatives if he is not searchable (coma).
* Affiliation to a social security system
* After an adapted preliminary medical examination

Exclusion Criteria:

* Post-traumatic meningeal hemorrhage
* Management time >48h with respect to bleeding
* Known neurodegenerative pathology (Alzheimer's, Parkinson's, etc.), Creutzfeldt-Jacob disease
* Pregnant woman
* Decision not to treat
* Refusal to participate in the study
* Adult patient protected by law
* Person deprived of administrative or judicial freedom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
median transit time (MTT) | 7 days
  median transit time (MTT) in seconds, on the perfusion scanner on 6 regions of the brain between D0 and D7 of the product perfusion

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Grenoble Hospital, Grenoble
  - Marseille Hospital, Marseille
  - Carole ICHAI, Nice

IPD SHARING:
Plan to Share IPD: No